CLINICAL TRIAL: NCT04985565
Title: Neoadjuvant Dietary Intervention in Intermediate Risk Prostate Cancer
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020-0673; NCI-2021-02022 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2020-0673 (Other: M D Anderson Cancer Center); P50CA140388 (NIH)
Record Dates: First submitted 2021-03-24; First posted 2021-08-02 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-09

CONDITIONS: Prostate Adenocarcinoma; Stage I Prostate Cancer AJCC v8; Stage II Prostate Cancer AJCC v8; Stage IIA Prostate Cancer AJCC v8; Stage IIB Prostate Cancer AJCC v8; Stage IIC Prostate Cancer AJCC v8; Stage IIIA Prostate Cancer AJCC v8
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Diet Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment (dietary intervention, radical prostatectomy) (Experimental): Patients participate in the Mediterranean diet for 6 days per week for 4 weeks before undergoing standard of care radical prostatectomy.
  Interventions: Other: Dietary Intervention; Procedure: Radical Prostatectomy

INTERVENTIONS:
Other: Dietary Intervention — Participate in Mediterranean diet
  Other Names: Dietary Modification; intervention, dietary; Nutrition Intervention; Nutrition Interventions; Nutritional Interventions
Procedure: Radical Prostatectomy — Undergo standard of care radical prostatectomy
  Other Names: Prostatovesiculectomy

SUMMARY:
This clinical trial studies the effects of a dietary intervention prior to surgery (neoadjuvant) in patients with intermediate risk prostate cancer. Changing your diet before surgery may help to improve overall health. Information from this study may help researchers better understand the influence of diet on the outcomes of patients with intermediate prostate cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine the feasibility of a neoadjuvant feeding study prior to radical prostatectomy in a racially diverse group of men diagnosed with intermediate risk prostate cancer, defined as the percentage of patients who enter the pre-intervention equilibration period and begin the dietary intervention.

SECONDARY OBJECTIVES:

I. Determine the tolerance of Mediterranean diet as defined by compliance with diet of 70% or greater total calories consumed during study period from the Mediterranean diet.

II. Determine the effects of controlled dietary interventions on metabolic parameters.

III. Determine the total number of potentially eligible patients who are approached by study coordinators and enter the equilibration period.

IV. Determine the effects of controlled dietary interventions on the fecal microbiome.

V. Create a well annotated bank of clinical data and samples, including but not limited to periprostatic fat, for use in future research and analysis.

VI. Examine the safety of controlled dietary interventions in patients with a diagnosis of prostate cancer.

VII. Determine changes in Cav-1-sphingolipid signature following Mediterranean diet consumption.

VIII. Compare Cav-1-sphingolipid levels following dietary interventions in with a separate cohort of men who do not undergo pre-operative dietary intervention.

OUTLINE:

Patients participate in the Mediterranean diet for 6 days per week for 4 weeks before undergoing standard of care radical prostatectomy.

After completion of study treatment, patients are followed up at 4-8 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed adenocarcinoma of the prostate that is localized based on prostate magnetic resonance imaging (MRI) and meets National Comprehensive Cancer Network (NCCN) intermediate risk criteria (as follows):

  * Clinical T2b-T2c or lower disease
  * Gleason Grade group 2 or 3 on biopsy
  * Prostate specific antigen (PSA) =< 20 ng/mL
  * Desires radical prostatectomy (open or robotic) for prostate cancer management and is a surgical candidate as determined by the treating urologic oncologist
* Adult men > 30 and < 75 years old (African American or non-Hispanic white)
* Meet one of the following criteria for overweight or obesity:

  * Body Mass Index (BMI) between 26 and 39
  * Waist circumference >= 40 inches
* Willingness to exclusively consume all the provided meals
* Willingness to comply with all study procedures and scheduled visits
* Reside in the greater Houston/outlying areas and/or willing to travel for study-related visits at MD Anderson

Exclusion Criteria:

* Major dietary restrictions or food allergies
* Food aversions or preferences that preclude following a Mediterranean diet, such as unwillingness to eat vegetables, grains, animal products or fish
* Medical contraindications to the intervention diet as determined by the treating physician
* Current self-reported smoker or heavy drinker (defined as >14 drinks per week) or current self-reported illicit drug use
* Prostate cancer that meets NCCN high and very high risk criteria (as follows):

  * pT3a or higher disease
  * Grade group 4 or 5 adenocarcinoma of prostate
  * PSA > 20ng/mL

Ages: 30 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2021-08-27 (Actual); Primary Completion 2025-10-20 (Estimated); Study Completion 2025-10-20 (Estimated)

PRIMARY OUTCOMES:
Feasibility of conducting a controlled feeding study in prostate cancer patients with intermediate risk disease | Up to 1 year from site initiation
  Feasibility is defined as >= 25% of patients who enter the equilibration period initiating the dietary intervention.

SECONDARY OUTCOMES:
Tolerance of Mediterranean diet | Up to 1 year
  Defined as compliance of 70% or greater total caloric intake consumed from the provided Mediterranean diet meals. Will estimate the number of patients that were compliant along with the 95% confidence intervals.
The effects of controlled dietary interventions on metabolic parameters | Up to 1 year
  As measured using metabolomics (Cav-1-signature score) and nuclear magnetic resonance (NMR) spectroscopy (using Nightingale platform). Paired t-test will be used to compare the metabolic parameters changes (pre- and post- dietary intervention) in untargeted mass spectrometry-based metabolite levels and NMR-based metabolite levels.
The effects of controlled dietary interventions on the fecal microbiome | Up to 1 year
  Exploratory analysis using microbiome core. Fecal microbiome samples will be summarized using alpha diversity, computed using the inverse Simpson index, which can then be compared across time points using a paired t-test.
Create a well annotated bank of clinical data and samples, including peri-prostatic fat, for use in future research and analysis | Up to 1 year
  Anticipate 100% participation in patients who enroll and complete diet intervention.
Examine the safety of controlled dietary interventions in patients with a diagnosis of prostate cancer percentage of severe adverse reactions in patients completing the diet. | Up to 1 year
Determine changes in Cav-1-sphingolipid signature following Mediterranean diet consumption | Up to 1 year
  Will compare the baseline Cav-1-signature score levels with the post-diet (day of surgery) levels using paired t-tests. This evaluation is exploratory in nature and will be used to guide power calculations for future studies.
Determine changes in Cav-1-sphingolipid signature following dietary intervention compared to a separate cohort with no intervention | Up to 1 year
  Will use a two-sample t-test to compare the levels of Cav-1-sphingolipid signature score in men who undergo a dietary intervention in this protocol with subjects enrolled under the separate protocol (protocol 2020-0828, "Diet, Biomarker, and Tissue Assessment in Intermediate Risk Prostate Cancer").

CONTACTS AND LOCATIONS:
Overall Officials: Justin R Gregg, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: M D Anderson Cancer Center — http://www.mdanderson.org

DOCUMENTS (1):
  • Informed Consent Form (2022-07-14): https://cdn.clinicaltrials.gov/large-docs/65/NCT04985565/ICF_000.pdf